CLINICAL TRIAL: NCT05040919
Title: Identification of Risk Factors for the Occurrence of High-grade Rhythm Disorders in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Identification of Risk Factors for the Occurrence of High-grade Rhythm Disorders in Patients With ST-segment Elevation Myocardial Infarction (STEMI)
Acronym: STEMI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: TIMSIT - Gevrey 2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Arrythmia -Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with an arrythmia: patient suffering from STEMI and presenting an arrythmia
  Interventions: Other: collection of medical and socio-demographic data
- without an arrythmia: patient suffering from STEMI and not presenting an arrythmia
  Interventions: Other: collection of medical and socio-demographic data

INTERVENTIONS:
Other: collection of medical and socio-demographic data — collection of medical and socio-demographic data

SUMMARY:
The goal of this study is to identify the risk factors for the occurrence of arrythmia in patient with stemi in prehospital management. We included 652 patients who presenting a STEMI from september 2017 to october 2020 and manage by physician in prehospital and bring to CHU of Dijon.

We analyse and compare the caracteristics of a group of STEMI patients who presenting an arrythmia to an other groupe of STEMI patient without arrythmia

ELIGIBILITY:
Inclusion Criteria:

> 18 years old, with STEMI, in prehospital patient, take by a medecine, bring to the CHU Dijon

Exclusion Criteria:

< 18 years old, without STEMI, no medical in prehospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every adult patient with a STEMI in prehospital, manage by a physician and bring to the CHU of Dijon
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
arrhythmia | at baseline
  arrhythmia during acute STEMI

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France